CLINICAL TRIAL: NCT05049434
Title: A Multi Center, Randomized, Single Blind, Assessor Blind, Matched Pair Design Clinical Study to Evaluate the Efficacy and Safety for Medicurtain® in Prevention of Adhesion After Endoscopic Sinus Surgery
Brief Title: Efficacy and Safety for Medicurtain® in Prevention of Adhesion After Endoscopic Sinus Surgery (Pivotal Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UMT2012-SP-MC-04
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Sinusitis; Tissue Adhesion, Surgery-Induced
Keywords: Medicurtain®; Sodium hyaluronate; Anti-adhesion barrier
MeSH Terms: conditions — Sinusitis; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Evaluator-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medicurtain® (Experimental): Treat GUARDIX-SG 5ml prefilled syringe after surgery
  Interventions: Device: Medicurtain®
- GUARDIX-SG® (Active Comparator): Treat Medicurtain® 5ml prefilled syringe after surgery
  Interventions: Device: GUARDIX-SG®

INTERVENTIONS:
Device: Medicurtain® — Medicurtain® 5ml prefilled syringe
  Arms: Medicurtain®
Device: GUARDIX-SG® — GUARDIX-SG® 5ml prefilled syringe
  Arms: GUARDIX-SG®

SUMMARY:
This clinical trial is to prove that the treatment group of Medicurtain® is non-inferior to the treatment group of Guardix-sol®, test equipment on adhesion after endoscopic sinus surgery, upon the aspects of adhesion prevention efficacy and safety.

DETAILED DESCRIPTION:
This clinical trial was conducted based on multi center, randomized, assessor blind, matched pair design, active-controlled clinical study. After signing consent and fulfilling the standards for selection/exclusion, test subjects went through required treatments following endoscopic surgery; subsequently, according to the order of registration after 2 to 3 days from the surgery, the subjects were applied with a medical device for the clinical test and a medical device for the control test to both of their nasal cavities based on randomization.

For procedures, bleeding was treated and prevented through packing, by soaking Merocel with saline solution following the ESS (Endoscopic sinus surgery) on subjects; and after 2 to 3 days (or upon discharge), it was to treat applied regions of the subjects with assigned medical device after confirming sufficient hemostasis by removing Merocel. Being matched pair active-controlled clinical study, this clinical trial was designed to treat a single subject with both medical devices for clinical test and control test where it was kept unknown which device would be assigned to which nasal cavity based on randomization until the procedure was actually performed. For the time and method of evaluation, observation and evaluation were allowed to be conducted based on the images through endoscopy when subjects visited at 1st, 2nd and 4th weeks following the treatment with medical device. The process of procedure was assured for an identical researcher to perform procedures in order to minimize the effect from the procedure method.

All endoscopic image records of test subjects were delivered by independent assessors, while information on medical device used for treatment was excluded; and independent assessors evaluated each image record according to the evaluation standards prescribed by this clinical trial.

Based on the determination of the researcher during and following the surgery, subjects were administered with 2nd or 3rd generation Cephalosporin Antibiotics. Following the surgery, subjects were instructed to use normal saline solution nasal spray 2 to 3 times a day on both nasal cavities by utilizing bulb-shape tube or syringe. In addition, subjects were also instructed to use intranasal steroid sprays.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at the age of between 19 and 69
2. Patients scheduled for surgery with chronic or relapsed sinusitis not responding to drug therapy (Verification to be made based on past clinical history, physical examination and radiography)
3. Patients with the discrepancy of Lund-MacKay CT scan scores on bilateral sinusitis less than 3
4. Patients who signed written consent after listening to the objective, method and effects of clinical trial
5. Patients available during the period of clinical trial

Exclusion Criteria:

1. Patients with sinusitis on only one nasal cavity
2. Patients with massive sinonasal polyposis
3. Patients with one or both middle turbinate removed, in addition to a history of endoscopic surgery or polyp operation
4. Patients with ongoing drug administration for asthma
5. Patients with immune disorders which may potentially hinder healing of the wounds including acquired immunodeficiency syndrome, cystofibroma, immotile cilia syndrome, neutropenia and immune globulin deficiency
6. Patients with immunosuppression or autoimmune disease
7. Patients with hypersensitivity reaction to Poloxamer and Hyaluronic acid
8. Patients who had surgery to treat extrasinus complication from rhinosinusitis
9. Patients with history of endoscopic sinus surgery for other than chronic or relapsed sinusitis, including cerebrospinal fluid (CSF) leak correction, orbital decompression and optic nerve decompression
10. Patients with significant liver or kidney diseases
11. Patients with setting agent administered or with hemostatic or lymph fluid disorders
12. Patients administered with oral or parenteral drugs for hypoglycemia
13. Patients with significant systematic disease
14. Patients with malignant tumor
15. Patients with infectious disease or suspected of potential problems during the course of healing surgical site (healing disorder)
16. Those who are pregnant or lactiferous
17. Women of childbearing age with plan for pregnancy during the clinical trial period
18. Those who participated in other clinical trials 30 days prior to the participation in this trial
19. In addition to the above, those who are subject to clinical findings where principal investigator or sub-investigator deem inadequate for this clinical trial based on medical judgment

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-03-03 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Difference between effective ratio (Pt=P00+P01) of medical device for clinical trial and effective ratio (Pc=P00+P10) of medical device for control test evaluated by independent assessor at the 4th week following the application of medical device | Week 4
  * P00: Ratio of study subjects without adhesion at the application site with medical devices for clinical trial and control test
  * P01: Ratio of study subjects without adhesion only at the application site with medical device for clinical trial
  * P10: Ratio of study subjects without adhesion only at the application site with medical device for control trial

SECONDARY OUTCOMES:
Ratio of study subjects without adhesion and extent of adhesion evaluated by independent assessor | follow up to 4weeks
  Adhesion is to be scored and recorded on the scale of 0 to 3 points, where the adhesion requiring treatments shall be scored at 2 points or higher. Independent assessor must be blind.
  * Standard for grading score of Synechia
  * Score 0: Synechia not visible
  * Score 1: One or a few synechia are visible, but clear hindrance obstructing sinus ventilation is not detected.
  * Score 2: Presence of Synechia obstructing sinus ventilation and drainage.
  * Score 3: Formation of complete scar between middle turbinate and lateral wall of nose.
Ratio of study subjects without adhesion and extent of adhesion evaluated by investigator | follow up to 4weeks
  Adhesion is to be scored and recorded on the scale of 0 to 3 points, where the adhesion requiring treatments shall be scored at 2 points or higher. Investigator is open-state.
Presence of adhesion (decomposition or dissolution) requiring treatments at 4th week | follow up to 4weeks
  Rate of patient who received 2 or more point in the adhesion assessment with medical devices for clinical trial or control test.
Ratio of study subjects without edema and the extent of edema evaluated at each visit | follow up to 4weeks
  Edema is to be score and record at the scale of 0 to 3 points, depending on the extensiveness where the case requiring treatments for edema with steroids shall be scored at 2 points or higher.
  * Standard for grading score of Edema
  * Score 0: Mucous membrane edema not visible
  * Score 1: Mild mucous membrane edema without extinction of ethmoid sinus
  * Score 2: Serious mucous membrane edema with extinction of most ethmoid sinus
  * Score 3: Parenchymatous polyposis
Presence of edema requiring treatment evaluated at each visit (Only the cases using oral steroid not for prevention purpose but for treatment purpose) | follow up to 4weeks
  Rate of patient who received 2 or more point in the edema assessment with medical devices for clinical trial or control test.
Ratio of study subjects without local infection and extent of local infection evaluated at each visit | follow up to 4weeks
  Infection is to be scored and recorded at the scale of 0 to 2 points where the case requiring treatments for infection shall be scored at 2 points.
  * Standard for grading score of Infection
  * Score 0: Proof of infection not visible
  * Score 1: Drainage of mild mucopurulent
  * Score 2: Drainage of lumpy mucopurulent accompanying parenchymatous infection
Presence of infection requiring treatment evaluated at each visit (Only the cases using antibiotics not for prevention purpose but for treatment purpose) | follow up to 4weeks
  Rate of patient who received 2 or more point in the infection assessment with medical devices for clinical trial or control test.

OTHER OUTCOMES:
The incidence rate of adverse events (AEs) | follow up to 4 weeks
  Safety and tolerability by collecting AEs

CONTACTS AND LOCATIONS:
Overall Officials: Heung-Man Lee, MD, Principal Investigator — Korea University, Guro Hospital 148 Gurodong-ro, Guro-gu, Seoul; Kyung-su Kim, MD, Principal Investigator — Gangnam Severance Hospital Yonsei University, 146-92 Dogok-dong, Gangnam-gu, Seoul
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No